CLINICAL TRIAL: NCT02471989
Title: Randomized Controlled Study of Low-FODMAP Diet in Patients With GERD Refractory to Protons Pump Inhibitors
Brief Title: FODMAPs and Refractory GERD
Acronym: EFFORR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2015/02
Record Dates: First submitted 2015-06-05; First posted 2015-06-15 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Gastro-esophageal Reflux Disease (GERD)
Keywords: FODMAP; Diet; pH-impedance monitoring
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-FODMAP diet (Experimental): FOS in diet
  Interventions: Dietary Supplement: Low-FODMAP diet
- Classical GERD diet (Active Comparator): avoid fatty meals, head of bed elevation...
  Interventions: Dietary Supplement: GERD diet

INTERVENTIONS:
Dietary Supplement: Low-FODMAP diet
  Arms: Low-FODMAP diet
Dietary Supplement: GERD diet
  Arms: Classical GERD diet

SUMMARY:
The aim of this study is to determine the effects of a low Fermentescible Oligosaccharides Disaccharides Monosaccharides and Polyols (FODMAP) diet in patients with documented refractory GERD on proton pump inhibitor (PPI) therapy.

DETAILED DESCRIPTION:
Colonic fermentation has been shown to influence oeso-gastric motility : increased gastric relaxation, increased rate of lower esophageal sphincter relaxation. Experimental increased colonic fermentation (FOS in diet) increase the occurrence of reflux events in patients with GERD. The aim of this study is to compare the low-FODMAP diet and classical GERD dietary recommendations (avoid fatty meals, head of bed elevation etc..) in patients with refractory GERD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Affiliation to French Social Security
* Informed written consent
* RDQ score > 3
* Abnormal pH-impedance monitoring on PPI twice daily (since 3 months) according to normal values published by Zerbib et al (CGH 2013)

Exclusion Criteria:

* Pregnancy or breast feeding
* Women of childbearing potential without an effective method of contraception
* Person under guardianship
* History of thoracic of abdominal surgery (excepted appendectomy and cholecystectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with clinical remission as defined by a RDQ score ≤ 3 | at Week 4 of diet

SECONDARY OUTCOMES:
Between-group comparison of efficacy | at Week 4 of diet
  This measure is a composite with :
  * Reflux Disease Questionnaire (RDQ) scores
  * Francis Irritable Bowel Syndrome (IBS) score
  * Quality of life (GIQLI) score
  * and reflux parameter on pH-impedance monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Frank ZERBIB, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (6):
- France (6):
  - Hépato-Gastroentérologie et oncologie digestive,, Bordeaux
  - Gastroentérologie, Colombes
  - Explorations fonctionnelles, Lyon
  - Gastroentérologie, Nantes
  - Explorations fonctionnelles Digestives, Rennes
  - Gastroentérologie, Rouen